CLINICAL TRIAL: NCT05136612
Title: Investigation Of The Effects Of Upper Extremity Robotic Rehabilitation On Upper Extremity Functions And Gait Parameters in Individuals With Cerebral Palsy
Brief Title: The Effects Of Upper Extremity Robotic Rehabilitation On Upper Extremity Functions And Gait Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Mustafa Burak, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021 -591
Record Dates: First submitted 2021-10-27; First posted 2021-11-29 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Individuals with CP will be assigned to group 1 or group 2 by simple randomization using the "Research Randomizer" program (https://www.randomizer.org/) prior to treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control grup (Experimental): conventional physiotherapy
  Interventions: Other: conventional physiothrapy
- intervention group (Experimental): Armeo spring robotic rehabilitation
  Interventions: Other: conventional physiothrapy; Other: robotic rehabilitation

INTERVENTIONS:
Other: conventional physiothrapy — Conventional physiotherapy program will be applied to the control group for 6 weeks, 3 days a week, 45 minutes a day. Strengthening, dynamic stretching, coordination and balance exercises and functional exercises for upper and lower extremities will be applied in this treatment program.
Other: robotic rehabilitation — The study group will be included in the rehabilitation program with the Hocoma brand Armeo Spring pediatric upper extremity robot for 30 minutes a day, 3 days a week, for 6 weeks at hospital. Armeo spring robot enables the individual to perform active movement by carrying the weight of the upper extremity of children who have active movement in their upper extremities but do not have enough strength to overcome gravity with their upper extremities. The individual is actively involved in the study during the study. With the adjustments made, it becomes suitable for use for right and left extremities. In the process of working; The games named High Flyer, Frisbee, Balloons, Goalkepper, Save the Monster, Fishing, Helicopter Rescue, which are included in the Armeo Spring robot and created to increase shoulder, elbow and wrist movements, will be used.
  Arms: intervention group

SUMMARY:
Cerebral Palsy is defined as the cause of movement and posture disorders and activity limitation that develops in the fetal or infant brain that has not yet completed its development. When the literature is examined, although upper extremity and lower extremity involvements are common in individuals with hemiparetic CP, treatment programs are mostly aimed at the lower extremities. However, studies report that the upper extremity is more severely affected than the lower extremities in individuals with hemiparetic CP and that upper extremity functions have an effect on walking. Although different treatment methods have positive effects, their superiority over each other cannot be clearly reported. In this case, new intervention strategies based on sound methodological and scientific foundations are needed. At this point, virtual reality applications and robotic rehabilitation programs have started to play an important role in CP rehabilitation along with current developments in technology-assisted rehabilitation. Robotic devices provide visual, auditory and sensory inputs, making the process fun, while making the individual active in the treatment. It also enables the child to achieve goal-directed movements in children with motor disabilities. Various gait problems are seen in individuals with CP. Therefore, although lower extremity movements during walking have been well analyzed in the literature, upper extremity functions and especially arm movements during walking have received less attention. Although human gait is perceived as a situation that concerns only the lower extremities, it actually includes the coordinated movements of all four extremities. Individuals with hemiplegic CP usually have a markedly deviated arm position and reduced arm movement. This situation also affects the gait and balance of individuals with hemiparetic CP. Individuals change their upper extremity kinematics while increasing their walking speed to optimize gait and increase balance. In the light of this information, practices aimed at improving upper extremity movement and function should be included in the rehabilitation program of patients with hemiparetic CP, considering a holistic approach. Considering all these, we thought that if we increase the functions of the upper extremities, we can improve walking, and we planned this study.

DETAILED DESCRIPTION:
Cerebral Palsy is defined as the cause of movement and posture disorders and activity limitation that develops in the fetal or infant brain that has not yet completed its development. Although CP is the most common physical disorder in childhood, its incidence varies between 1.7-2 people per 1000 live births in developed countries. Although the impairments seen in CP are not progressive, as individuals with CP get older, their current motor function declines dramatically and their independence decreases or disappears as a result. These neurodevelopmental disorders are classified as hemiplegic, diplegic and quadriplegic according to the anatomically affected body parts. Along with motor damage, epilepsy, cognitive disorders, behavioral disorders, visual-hearing losses and sensory disorders can be seen in children with CP. In addition, upper extremity involvement is quite common in individuals with CP. Although upper extremity and lower extremity involvement are common in individuals with hemiparetic CP, treatment programs are mostly aimed at the lower extremities. However, studies report that the upper extremity is more severely affected than the lower extremities in individuals with hemiparetic CP and that upper extremity functions have an effect on walking . Although human gait is perceived as a situation that concerns only the lower extremities, it actually includes the coordinated movements of all four extremities. In a study, it was reported that it is beneficial to encourage arm movements during gait rehabilitation. It has been reported that although individuals with hemiparetic CP gain walking skills, they lag behind their peers in terms of upper extremity functions. This makes upper extremity rehabilitation important. There are various treatment modalities aimed at eliminating upper extremity dysfunction and reducing activity limitations. These; neurodevelopmental treatment approaches, orthoses, forced restrictive movement therapy, virtual reality and robotic rehabilitation applications. Although the different treatment methods have positive effects, their superiority to each other cannot be reported definitively. In this case, new intervention strategies based on sound methodological and scientific foundations are needed.

With the development of technology, the interest in robotic rehabilitation has also increased. The first study examining upper extremity robotic rehabilitation in CP was conducted in 2008. In this study, it was reported that robotic rehabilitation has positive effects on upper extremity motor functions and the use of upper extremities in daily living activities. In a thesis study conducted in our country, conventional physiotherapy and robotic rehabilitation were compared and it was concluded that hand skills improved in both groups, but the increase in the group receiving robotic rehabilitation was statistically significant. In the literature review, it was seen that studies on upper extremity robotic rehabilitation were few and their effects on gait parameters were not examined. In this context, it is thought that in our study, the effects of upper extremity robotic rehabilitation on upper extremity functions and gait parameters will be examined and it will contribute to the literature.

Method: This study was conducted to examine the effects of upper extremity robotic rehabilitation on upper extremity functions and gait parameters in individuals with hemiparetic CP; It is a prospective, randomized controlled, single-blind study. The study will be carried out in a single-blind manner, and the evaluator will not know which group the individual is in. 30 individuals with spastic hemiparetic CP, aged between 6-18 years, will be included in our study. The parents of each individual will be informed about the study and will read and sign the consent form stating that they voluntarily participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* The clinical type is spastic hemiparetic CP.
* Upper extremity spasticity value between 0 and 3 according to Modified Ashworth.
* To have the cognitive level to understand simple instructions.
* It is largely the absence of auditory and visual loss.

Exclusion Criteria:

* not volunteering to participate in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Data Form | Before starting treatment
  Information such as gender, age, clinical type, extremity involvement, dominant extremity, birth weight, assistive devices used of the cases will be recorded in the prepared sociodemographic data form.
Joint Range of Motion (ROM) Measurement | Before starting treatment
  Individuals' ROM degrees will be evaluated before and after the treatment using a universal goniometer in the supine position. Individuals' shoulder flexion, abduction, internal and external rotation, elbow and wrist flexion and extension painless active ROM measurements will be evaluated and recorded bilaterally.
Functional Independence Measure for Children (WeeFIM) | Before starting treatment
  The WeeFIM is derived from the Functional Independence Measure (FIM) and includes 18 items involving six functional subscalcs. It is used to detect the functional independence levels of children and changes in time-dependent functions.
Pediatric Quality of Life Inventory | Before starting treatment
  The Pediatric Quality of Life Inventory (PedsQL™) is a modular instrument for measuring health-related quality of life dimensions in children and adolescents ages 2-18 years. The PedsQL™ 4.0 Generic Core Scales are multidimensional (physical, emotional, social, school/role functioning) child self-report and parent proxy report scales developed as a generic measure to be integrated with the PedsQL™ disease-specific modules.
The Jebsen Hand Function Test | Before starting treatment
  The Jebsen Hand Function Test (JHFT) was developed to provide a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. It has 7 items and takes approximately 15-45 minutes to administer.
  Item 1: Writing, Item 2: Card Turning, Item 3: Small Common Objects, Item 4: Simulated feeding, Item 5: Checkers, Item 6: Large Light Object, Item 7: Large Heavy Objects
ABILHAND-Kids | Before starting treatment
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. The ABILHAND-Kids questionnaire assesses manual ability as a test focused on the child's difficulty perceived by the child's parents.
  The questionnaire was developed using the Rasch measurement model which provides a method to convert the raw scores into a linear measure located on a unidimensional scale.
  ABILHAND-Kids has been calibrated in children with cerebral palsy according to the difficulty of children in performing manual activities as perceived by their parents.
The Quality of Upper Extremity Skills Test | Before starting treatment
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. There are 36 items that evaluate dissociated movements, grip, protective extension, and weight bearing.
Selective Control of the Upper Extremity Scale | Before starting treatment
  This test was developed to evaluate the selective motor control of the upper extremity. It is a very practical and useful video-based assessment tool that can be applied in less than 15 minutes. No special equipment is required other than a video camera. It offers the opportunity to evaluate the selective movements of the shoulder, elbow, forearm, wrist and fingers for both right and left extremities. The person administering the test passively shows the participant the movements they are asked to do. Then the participant is asked to actively perform the movement shown. While performing the participant movements; Head, trunk and other extremity movements are taken with a video camera to provide the opportunity to observe. The degree of selective motor control is determined as 0-3 points for each joint, depending on the person's ability to perform movements and their shape.
Trunk Control Measurement Scale | Before starting treatment
  The Trunk Control Measurement Scale (TCMS) was used to evaluate the trunk control of the individuals participating in the study. The TCMS includes 15 items that measure static and dynamic sitting balance, the two main components of trunk control. The Static Sitting Balance Scale (item 1-5) evaluates the ability to maintain a stable trunk posture during movements of the upper and lower extremities. The Dynamic Sitting Balance Scale (item 6-15) is divided into two subscales, the selective movement control scale and the dynamic reaching scale. The total score is between 0-58. A higher score indicates better performance.
4D Diers Formetic | Before starting treatment
  In this study, the newly developed 4D Diers Formetic movable spine and surface topography evaluation device will be used. This device is equipped with a digital network camera that allows measurements at a maximum frequency of up to 50 frames per second. The camera uses CMOS sensors with a resolution of 1280x1024 pixels. Thanks to these sensors and reflective markers, measurements are reconstructed in 3D. Thus, it allows real-time evaluation of posture and gait parameters. Evaluation is done without radiation and without contact.
Sociodemographic Data Form | After 6 weeks of treatment (treatment is 18 sessions)
  Information such as gender, age, clinical type, extremity involvement, dominant extremity, birth weight, assistive devices used of the cases will be recorded in the prepared sociodemographic data form.
Joint Range of Motion (ROM) Measurement | After 6 weeks of treatment (treatment is 18 sessions)
  Individuals' ROM degrees will be evaluated before and after the treatment using a universal goniometer in the supine position. Individuals' shoulder flexion, abduction, internal and external rotation, elbow and wrist flexion and extension painless active ROM measurements will be evaluated and recorded bilaterally.
Functional Independence Measure for Children (WeeFIM) | After 6 weeks of treatment (treatment is 18 sessions)
  The WeeFIM is derived from the Functional Independence Measure (FIM) and includes 18 items involving six functional subscalcs. It is used to detect the functional independence levels of children and changes in time-dependent functions.
Pediatric Quality of Life Inventory | After 6 weeks of treatment (treatment is 18 sessions)
  The Pediatric Quality of Life Inventory (PedsQL™) is a modular instrument for measuring health-related quality of life dimensions in children and adolescents ages 2-18 years. The PedsQL™ 4.0 Generic Core Scales are multidimensional (physical, emotional, social, school/role functioning) child self-report and parent proxy report scales developed as a generic measure to be integrated with the PedsQL™ disease-specific modules.
The Jebsen Hand Function Test | After 6 weeks of treatment (treatment is 18 sessions)
  The Jebsen Hand Function Test (JHFT) was developed to provide a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. It has 7 items and takes approximately 15-45 minutes to administer.
  Item 1: Writing, Item 2: Card Turning, Item 3: Small Common Objects, Item 4: Simulated feeding, Item 5: Checkers, Item 6: Large Light Object, Item 7: Large Heavy Objects
ABILHAND-Kids | After 6 weeks of treatment (treatment is 18 sessions)
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs, whatever the strategies involved. The ABILHAND-Kids questionnaire assesses manual ability as a test focused on the child's difficulty perceived by the child's parents.
  The questionnaire was developed using the Rasch measurement model which provides a method to convert the raw scores into a linear measure located on a unidimensional scale.
  ABILHAND-Kids has been calibrated in children with cerebral palsy according to the difficulty of children in performing manual activities as perceived by their parents.
The Quality of Upper Extremity Skills Test | After 6 weeks of treatment (treatment is 18 sessions)
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. There are 36 items that evaluate dissociated movements, grip, protective extension, and weight bearing.
Selective Control of the Upper Extremity Scale | After 6 weeks of treatment (treatment is 18 sessions)
  This test was developed to evaluate the selective motor control of the upper extremity. It is a very practical and useful video-based assessment tool that can be applied in less than 15 minutes. No special equipment is required other than a video camera. It offers the opportunity to evaluate the selective movements of the shoulder, elbow, forearm, wrist and fingers for both right and left extremities. The person administering the test passively shows the participant the movements they are asked to do. Then the participant is asked to actively perform the movement shown. While performing the participant movements; Head, trunk and other extremity movements are taken with a video camera to provide the opportunity to observe. The degree of selective motor control is determined as 0-3 points for each joint, depending on the person's ability to perform movements and their shape.
Trunk Control Measurement Scale | After 6 weeks of treatment (treatment is 18 sessions)
  The Trunk Control Measurement Scale (TCMS) was used to evaluate the trunk control of the individuals participating in the study. The TCMS includes 15 items that measure static and dynamic sitting balance, the two main components of trunk control. The Static Sitting Balance Scale (item 1-5) evaluates the ability to maintain a stable trunk posture during movements of the upper and lower extremities. The Dynamic Sitting Balance Scale (item 6-15) is divided into two subscales, the selective movement control scale and the dynamic reaching scale. The total score is between 0-58. A higher score indicates better performance.
4D Diers Formetic | After 6 weeks of treatment (treatment is 18 sessions)
  In this study, the newly developed 4D Diers Formetic movable spine and surface topography evaluation device will be used. This device is equipped with a digital network camera that allows measurements at a maximum frequency of up to 50 frames per second. The camera uses CMOS sensors with a resolution of 1280x1024 pixels. Thanks to these sensors and reflective markers, measurements are reconstructed in 3D. Thus, it allows real-time evaluation of posture and gait parameters. In the evaluation, the individual's single stance left, right single stance, stance phase right, stance right left and double stance will be recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa BURAK, Phd, Principal Investigator — bulentelbasan@gmail.com
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] El-Shamy SM. Efficacy of Armeo(R) Robotic Therapy Versus Conventional Therapy on Upper Limb Function in Children With Hemiplegic Cerebral Palsy. Am J Phys Med Rehabil. 2018 Mar;97(3):164-169. doi: 10.1097/PHM.0000000000000852. PMID 29059068
- [Background] Dixit S, Tedla JS. Effectiveness of robotics in improving upper extremity functions among people with neurological dysfunction: a systematic review. Int J Neurosci. 2019 Apr;129(4):369-383. doi: 10.1080/00207454.2018.1536051. Epub 2018 Nov 22. PMID 30311823